CLINICAL TRIAL: NCT02784132
Title: Video Diversion Improves the Success Rate of Fundoscopic Examination in Children: a Prospective Multi-clinic, Multi-practitioner, Randomized Controlled Trial
Brief Title: Video Diversion Improves Success Rate of Fundoscopic Examination in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: None | Purpose: Diagnostic
Other Study IDs: H12-02053
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2016-05

CONDITIONS: Fundoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Study Arm A (Other): Right eye examined first with video diversion then left eye examined without video diversion
  Interventions: Other: Video diversion
- Study Arm B (Other): Right eye examined first without video diversion then left eye examined with video diversion
  Interventions: Other: Video diversion
- Study Arm C (Other): Left eye examined first with video diversion then right eye examined without video diversion
  Interventions: Other: Video diversion
- Study Arm D (Other): Left eye examined first without video diversion then right eye examined with video diversion
  Interventions: Other: Video diversion

INTERVENTIONS:
Other: Video diversion — The intervention is playing a video on a computer or iPad (using www.youtube.com) while performing fundoscopy.

SUMMARY:
Fundoscopy is an important component of the neurological examination as it can detect pathologies such as high intracranial pressure. However, the exam can be challenging in uncooperative children. This study looked at whether playing a video during eye examination, improves the success, duration and ease of pediatric fundoscopy.

DETAILED DESCRIPTION:
Fundoscopy is an important component of the neurological examination as it can detect pathologies such as high intracranial pressure. However, the exam can be challenging in uncooperative children. This study looked at whether playing a video during eye examination, improves the success, duration and ease of pediatric fundoscopy. The authors plan to recruit from 4 different clinical care settings for a total of 101 subjects. Success rate is defined as visualizing the optic disc within 60 seconds from commencement of fundoscopy. The ease of examination is determined by using a 10 point likert scale.

ELIGIBILITY:
Inclusion Criteria:

* patient aged 1 to 4 years of age (inclusive) with 2 examinable eyes

Exclusion Criteria:

* Patients who were blind, younger than 1 year of age, or older than 4 years of age

Ages: 1 Year to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Success rate of visualizing the optic disc within 60 seconds | 60 second

SECONDARY OUTCOMES:
Time required to visualize the optic disc | 60 seconds
Ease of performing fundoscopy | 60 seconds

CONTACTS AND LOCATIONS:
Overall Officials: Ash Singhal, Dr., Principal Investigator — The University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang MMH, Singhal A, Hengel AR, Kerr JM, St-Pierre GH, George S, Muir K, Thiessen P, Enarson P. Video Diversion Improves Success Rate of Fundoscopic Examination in Children: A Prospective Randomized Controlled Trial. Pediatr Neurol. 2018 Jun;83:32-37. doi: 10.1016/j.pediatrneurol.2017.09.008. Epub 2017 Sep 14. PMID 29681489